CLINICAL TRIAL: NCT03701269
Title: Long-term Radiographic and Clinic Surgical Outcomes of Scaphoid Proximal Pole Fracture Nonunion
Brief Title: Long-term Surgical Outcomes of Scaphoid Proximal Pole Fracture Nonunion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018-08-010AC
Record Dates: First submitted 2018-09-26; First posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Orthopedic
Keywords: Fracture
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The treatment for scaphoid proximal pole nonunion remains challenging due to the poor vascularity in the proximal pole fragment, associated SL injury and the technique of fixation. Vascularized bone grafts and non-vascularized iliac bone graft have been used in patients with scaphoid proximal pole nonunion, but the indication has not been well clarified. Alternatively, we have been treating such patients with vascularized bone graft , or non-vascularized bone graft with screw or k-wire fixation with considerable success. The purpose of this study is to evaluate and analyze retrospectively the surgical efficacy of our procedure.

DETAILED DESCRIPTION:
Scaphoid nonunion are common and operative treatment with bone graft was reported to have good result. However, the treatment for proximal pole nonunion remains controversial. There are some patterns of pathoanatomy combined with scaphoid fracture, like SL ligament tears, which could not be easily identified or treated initially. The proximal pole nonunion was near SL joint. Therefore, proximal pole nonunion may result in DISI instability. Furthermore, proximal pole nonunion was identified as a poor prognostic factor in scaphoid nonunion.

In the past 10 years, we have some different technique, like VBG, arthroscopic bone graft to achieve good results. Some studies revealed that significantly better SL stability was achieved with ARASL. We also used ARASL with BG to improve proximal pole union. However, it is not clear which method would be appropriate for proximal pole nonunion. We retrospectively investigated the functional outcome and radiological results after at least 2-year follow-up to clarify the surgical efficacy of these procedures.

ELIGIBILITY:
Inclusion Criteria:

* (1) chronic nonunion (wrist pain for more than 3 months after injury) as defined by preoperative radiographs; and (2) combined positive SL instability measured by intraoperative arthroscopy exam test; (3) Grade I SNAC.

Exclusion Criteria:

* (1) skeletally immature patients; (2) previous wrist trauma or surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Using arthroscopic or open fixation combined with bone graft surgery for proximal pole scaphoid nonunion
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-08-14 (Actual); Primary Completion 2019-08-13 (Estimated); Study Completion 2019-08-13 (Estimated)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand (DASH) score | averaged 2 years
  30-item disability/symptom scale, scored 0 (no disability) to 100

SECONDARY OUTCOMES:
Radiographic examination | averaged 2 years
  The union was defined as trabecular bridging across the fracture site

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Pan Wang, M.D.,ph.D, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan